CLINICAL TRIAL: NCT05232188
Title: The Effect of Renal Access Sheath Size Used During Percutaneous Nephrolithotomy on Postoperative Renal Functions
Brief Title: Effect of Renal Access Sheath on Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NoyanOzluPCNL
Record Dates: First submitted 2021-11-25; First posted 2022-02-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Kidney Function Tests; Treatment Outcome
Keywords: Percutaneous nephrolithotomy; Amplatz sheath
MeSH Terms: interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22French (Fr) (Experimental): After renal access, dilatation is provided up to 22Fr with a dilatator set, and fragmentation is started with a 19Fr nephroscope.
  Interventions: Procedure: Percutaneous nephrolithotomy
- 28F (Experimental): After renal access, dilatation is provided up to 28Fr with a dilatator set, and fragmentation is started with a 25Fr nephroscope.
  Interventions: Procedure: Percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy — percutaneous nephrolithotomy surgery, 22F amplatz sheath is used in one group, while 28F amplatz sheath is used in the other group.

SUMMARY:
Patients will be randomly divided into two groups in order to evaluate the effect of the size of the access sheath (Amplatz) used in the Percutaneous Nephrolithotomy (PCNL) operation on kidney functions. After dilatation, 22French (Fr) Amplatz sheath will be placed in the first group, while 28Fr Amplatz sheath will be placed in the second group.

The functional difference will be evaluated with preoperative and postoperative 3rd-month kidney scintigraphies (diethylenetriamine pentaacetic acid (DTPA) and technetium-99m dimercaptosuccinic acid (DMSA). In addition, Kidney Injury Molecule-1 (KIM-1) levels will be measured in the urine in order to be a predictor of functional loss in the early period.

DETAILED DESCRIPTION:
PCNL has been applied for the last 30 years as the primary and most effective treatment method in patients with kidney stones of 2 cm or larger. The primary purpose of the operation is to ensure stone-freeness. Another aim is to keep the damage to kidney functions to a minimum, thanks to the endoscopic intervention. In this respect, PCNL is superior to open surgery and reduces morbidity.

Renal access, dilatation, and fragmentation are the 3 important stages of the operation, and access and dilation significantly affect the final results of PCNL. The size of the access sheath used as a result of dilation determines the size of the tract where the endoscopic intervention will be made, and not only affects the postoperative results and success but also determines the factors that may affect the kidney functions such as bleeding and loss of parenchyma in the kidney.

There are studies showing that less bleeding, shorter hospital stay, and better postoperative pain control are achieved with the reduction of access sheath size. In addition to conventional PCNL, methods such as mini PCNL, micro PCNL, ultra-mini PCNL, and tubeless PCNL, where the diameter of the access sheath and endoscope are gradually decreasing, both increase success and reduce morbidity.

In our study, in order to examine the postoperative functional results of 22 Fr and 28 Fr accessory sheath size;

* For the early period, the change in KIM-1 values, a validated biomarker in acute kidney injury, measured on the preoperative and postoperative day 1 will be proportioned between the groups,
* For the late period, we aimed to compare the kidney functions in the mid-long term by proportioning the DMSA and DTPA values at the preoperative and postoperative 3rd month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2-3 cm kidney stones
* Patients with an American Society of Anesthesiologists ≤2 score
* BMI: Patients between 20 and 35 kg/m2

Exclusion Criteria:

* Patients with preoperative renal failure
* Patients with multiple access
* Patients undergone renal transplantation
* Patients with renal anomalies (horseshoe kidney, solitary kidney, double collecting system, etc.)
* Patients with history of open kidney stones surgery and/or PCNL history
* Patients who cannot be stone-free in the postoperative period (fragments >4 mm in imaging) and require additional treatment intervention
* Patients with bleeding disorders
* Pregnant patients
* Patients with complete staghorn stones
* Patients with bilateral obstructive stones
* Patients with active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Differential function changes | 3 months
  Differential function changes in the operated kidney in postoperative DMSA and DTPA
Newly developed scar | 3 months
  Presence of newly developed scar in DMSA
KIM-1 | 24 hours
  Change in urinary KIM-1 levels

SECONDARY OUTCOMES:
Creatinine | 24 hours
  Postoperative changes in creatinine
Glomerular filtration rate | 24 hours
  Postoperative changes in glomerular filtration rate
Stone-free rate | 24 hours
  Postoperative stone-free rates
Complications | 30 days
  Complications according to Clavian grading

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)